CLINICAL TRIAL: NCT05744518
Title: Monitoring Response to Neoadjuvant Chemotherapy in Breast Cancer Using Ultrafast Dynamic Contrasted-Enhancement Magnetic Resonance Imaging
Brief Title: Monitoring Response to Neoadjuvant Chemotherapy in Breast Cancer Using Ultrafast DCE-MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yajia Gu, MD, Director, Head of Radiology, Principal Investigator, Clinical Professor, Fudan University
Other Study IDs: MR-01
Record Dates: First submitted 2023-01-28; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Response monitoring — Other: Response monitoring (no intervention)

SUMMARY:
The study will assess whether changes in kinetic parameters of tumor and peritumoral vasculature using ultrafast dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) during neoadjuvant chemotherapy (NAC) are predictive of pathologic complete response (pCR) in patients with breast cancer appropriate for NAC. pCR is defined as having no residual invasive breast cancer or ductal carcinoma in situ.

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Age 18 years or older;
3. Diagnosis of invasive breast cancer by ultrasound guided biopsy;

3. Planed for receiving neoadjuvant chemotherapy (NAC) 4. Planned definitive breast surgery following completion of NAC.

Exclusion Criteria:

1. Stage IV breast cancer;
2. Previous ipsilateral breast cancer;
3. Previous treatment (chemotherapy or radiation) to involved breast;
4. Medically unstable;
5. Pregnant or nursing.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Eligible female breast cancer patients receiving NAC at Fudan University Shanghai Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-01-03 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Complete Pathologic Response (pCR) | 6 Months Post Surgery
  The primary aim of this feasibility study is to determine whether ultrafast dynamic contrasted-enhancement magnetic resonance imaging (DCE-MRI) at baseline prior to first cycle neoadjuvant chemotherapy (NAC), after first cycle NAC, and prior to second cycle NAC can accurately predict complete pathologic response (pCR) in women with breast cancer.

SECONDARY OUTCOMES:
Image Quality | 6 Months Post Surgery
  The second aim of this feasibility study is to determine whether ultrafast dynamic contrasted-enhancement magnetic resonance imaging (DCE-MRI) can provide the relatively high resolution, high contrast-noise ration, and good contrast with ultrafast DCE-MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided